CLINICAL TRIAL: NCT02732483
Title: Role of Hemostatic Powder (Endo-clotTM) in Success and Prevention of Bleeding Within Gastric Cancer Patients With Bleeding
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 4-2016-0031
Record Dates: First submitted 2016-03-27; First posted 2016-04-08 (Estimated); Last update posted 2016-04-08 (Estimated); Status verified 2016-04

CONDITIONS: Bleeding at Gastric Cancer
Keywords: gastric cancer; bleeding; gastrointestinal hemorrhage
MeSH Terms: conditions — Stomach Neoplasms; Hemorrhage; Gastrointestinal Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Endo-Clot(TM) (Experimental)
  Interventions: Drug: Endo-Clot(TM)

INTERVENTIONS:
Drug: Endo-Clot(TM) — The patients agreed in this study, bleeding control will going to be done with Endo-Clot(TM)

SUMMARY:
Gastrointestinal(GI) hemorrhage related with gastric cancer is prevalent in advanced cases mostly. As endoscopic hemostatic methods such as argon plasma ablation (APC) had developed, controlling GI hemorrhage in gastric cancer is much easier these days. but re-bleeding rate is still high, even after successful hemostasis with APC or electrical coagulation. Furthermore patients who were experienced re-bleeding are expected poorer survival outcomes than those who are not. So excellent bleeding control in gastric cancer is most important in GI hemorrhage of gastric cancer.

Recently developed hemostatic powder [Endo-Clot(TM)] is easy to use and have proven its usefulness in GI hemorrhage in peptic ulcer diseases. So in this study, investigator will try to find out feasibility & safety of Endo-Clot(TM) in GI hemorrhage in gastric cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age over 19 and less 80 yeas old
* Gastric cancer was diagnosed with biopsy and/or computed tomography
* Endoscopic hemostasis is needed upto GI hemorrhage
* Endoscopic examination is available in 24hours
* ECOG performance status(PS) <2

Exclusion Criteria:

* Double primary caner
* Hypersensitivity of hemostatic power[Endo-Clot(TM)]
* Variceal bleeding or benign gastric ulcer bleeding
* Hemodynamically unstable with low systolic BP<90mmHg and/or tachycardia PR>120bpm
* endoscopic hemostasis within 7 days before screening
* Contraindication for endoscopic examination
* Pregnant
* Breast feeding
* bleeding tendency with low platelet count <50,000 /mm^3 and/or INR>2
* Bacterial infection with needs for antibiotics therapy
* Unavailable to discontinue anti-coagulation agent for 3days
* Vascular shunt
* Cardiovascular and/or pulmonary diseases
* Active hepatitis or severe liver diseases
* Renal dysfunction
* Bone marrow dysfunction
* Neurologic deficit and/or psychotic feature
* Unavailable informed consent

Ages: 19 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2016-04; Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Rebleeding rate | within 30 days
  Proportion of patients who are experience rebleeding events after hemostasis within 30 days expected to be lower than 10 %.
  Definition rebleeding events 1. Overt symptoms of GI bleeding(such as hematemesis, melena) and/or Hemoglobin down more than 2g/dl compared to Hemoglobin level which were checked just after procedure.

SECONDARY OUTCOMES:
Success of bleeding control rate | within 2 weeks and 4 weeks
  Proportion of patients who are experience successful hemostasis is expected to be higher than 80 %applying Endo-Clot™, Rebleeding rate in 3days, rate of additional intervention other than initial endoscopic hemostasis, Mortalities
Rebleeding rate | in 3 days
  Proportion of patients experience rebleeding events after hemostasis within 3 days expected to be lower than 5 %. Definition of Rebleeding rate in 3days 1. Overt symptoms of GI bleeding(such as hematemesis, melena) and/or Hemoglobin down more than 2g/dl compared to Hemoglobin level which were checked just after procedure.
Rate of additional intervention other than initial endoscopic hemostasis | within 2 weeks to 4 weeks
  Definition of Successful hemostasis; controlled bleeding vessel in 5 minute after applying Endo-Clot™
Mortalities | within 2 weeks to 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Internal Medicine,, Seoul, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
no plan to share data

REFERENCES:
- [Result] Thrumurthy SG, Chaudry MA, Hochhauser D, Mughal M. The diagnosis and management of gastric cancer. BMJ. 2013 Nov 4;347:f6367. doi: 10.1136/bmj.f6367. No abstract available. PMID 24191271
- [Result] Chaw CL, Niblock PG, Chaw CS, Adamson DJ. The role of palliative radiotherapy for haemostasis in unresectable gastric cancer: a single-institution experience. Ecancermedicalscience. 2014 Jan 10;8:384. doi: 10.3332/ecancer.2014.384. eCollection 2014. PMID 24482669
- [Result] Lee HJ, Yang HK, Ahn YO. Gastric cancer in Korea. Gastric Cancer. 2002;5(3):177-82. doi: 10.1007/s101200200031. No abstract available. PMID 12378346
- [Result] Isobe Y, Nashimoto A, Akazawa K, Oda I, Hayashi K, Miyashiro I, Katai H, Tsujitani S, Kodera Y, Seto Y, Kaminishi M. Gastric cancer treatment in Japan: 2008 annual report of the JGCA nationwide registry. Gastric Cancer. 2011 Oct;14(4):301-16. doi: 10.1007/s10120-011-0085-6. Epub 2011 Sep 7. PMID 21894577
- [Result] Lasithiotakis K, Antoniou SA, Antoniou GA, Kaklamanos I, Zoras O. Gastrectomy for stage IV gastric cancer. a systematic review and meta-analysis. Anticancer Res. 2014 May;34(5):2079-85. PMID 24778009
- [Result] Romera Barba E, Castaner Ramon-Llin J, Sanchez Perez A, Garcia Marcilla JA, Vazquez Rojas JL. Transcatheter arterial embolization in the management of acute bleeding from advanced gastric cancer. Cir Esp. 2014 Aug-Sep;92(7):492-4. doi: 10.1016/j.ciresp.2013.11.004. Epub 2013 Dec 27. No abstract available. English, Spanish. PMID 24378191
- [Result] Sheibani S, Kim JJ, Chen B, Park S, Saberi B, Keyashian K, Buxbaum J, Laine L. Natural history of acute upper GI bleeding due to tumours: short-term success and long-term recurrence with or without endoscopic therapy. Aliment Pharmacol Ther. 2013 Jul;38(2):144-50. doi: 10.1111/apt.12347. Epub 2013 May 28. PMID 23710797
- [Result] Kim YI, Choi IJ, Cho SJ, Lee JY, Kim CG, Kim MJ, Ryu KW, Kim YW, Park YI. Outcome of endoscopic therapy for cancer bleeding in patients with unresectable gastric cancer. J Gastroenterol Hepatol. 2013 Sep;28(9):1489-95. doi: 10.1111/jgh.12262. PMID 23662891
- [Result] Kim MM, Rana V, Janjan NA, Das P, Phan AT, Delclos ME, Mansfield PF, Ajani JA, Crane CH, Krishnan S. Clinical benefit of palliative radiation therapy in advanced gastric cancer. Acta Oncol. 2008;47(3):421-7. doi: 10.1080/02841860701621233. PMID 17899453
- [Result] Hashimoto K, Mayahara H, Takashima A, Nakajima TE, Kato K, Hamaguchi T, Ito Y, Yamada Y, Kagami Y, Itami J, Shimada Y. Palliative radiation therapy for hemorrhage of unresectable gastric cancer: a single institute experience. J Cancer Res Clin Oncol. 2009 Aug;135(8):1117-23. doi: 10.1007/s00432-009-0553-0. Epub 2009 Feb 10. PMID 19205735
- [Result] Asakura H, Hashimoto T, Harada H, Mizumoto M, Furutani K, Hasuike N, Matsuoka M, Ono H, Boku N, Nishimura T. Palliative radiotherapy for bleeding from advanced gastric cancer: is a schedule of 30 Gy in 10 fractions adequate? J Cancer Res Clin Oncol. 2011 Jan;137(1):125-30. doi: 10.1007/s00432-010-0866-z. Epub 2010 Mar 25. PMID 20336314
- [Result] Tey J, Choo BA, Leong CN, Loy EY, Wong LC, Lim K, Lu JJ, Koh WY. Clinical outcome of palliative radiotherapy for locally advanced symptomatic gastric cancer in the modern era. Medicine (Baltimore). 2014 Nov;93(22):e118. doi: 10.1097/MD.0000000000000118. PMID 25396330
- [Result] Ono S, Ono M, Nakagawa M, Shimizu Y, Kato M, Sakamoto N. Delayed bleeding and hemorrhage of mucosal defects after gastric endoscopic submucosal dissection on second-look endoscopy. Gastric Cancer. 2016 Apr;19(2):561-567. doi: 10.1007/s10120-015-0507-y. Epub 2015 Jun 19. PMID 26089283
- [Result] Kim SB, Lee SH, Kim KO, Jang BI, Kim TN, Jeon SW, Kwon JG, Kim EY, Jung JT, Park KS, Cho KB, Kim ES, Kim HJ, Park CK, Park JB, Yang CH. Risk Factors Associated with Rebleeding in Patients with High Risk Peptic Ulcer Bleeding: Focusing on the Role of Second Look Endoscopy. Dig Dis Sci. 2016 Feb;61(2):517-22. doi: 10.1007/s10620-015-3846-y. Epub 2015 Aug 22. PMID 26297133
- [Result] Bustamante-Balen M, Plume G. Role of hemostatic powders in the endoscopic management of gastrointestinal bleeding. World J Gastrointest Pathophysiol. 2014 Aug 15;5(3):284-92. doi: 10.4291/wjgp.v5.i3.284. PMID 25133029
- [Result] Huang R, Pan Y, Hui N, Guo X, Zhang L, Wang X, Zhang R, Luo H, Zhou X, Tao Q, Liu Z, Wu K. Polysaccharide hemostatic system for hemostasis management in colorectal endoscopic mucosal resection. Dig Endosc. 2014 Jan;26(1):63-8. doi: 10.1111/den.12054. Epub 2013 Mar 31. PMID 23551344